CLINICAL TRIAL: NCT05965050
Title: Effect Of Myofascial Release Technique With Ultrasound Therapy in Adults With Nonspecific Low Back Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DPT/Batch-Fall18/541
Record Dates: First submitted 2023-03-18; First posted 2023-07-28 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Ultrasonic Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myofascial Release Technique (Other): myofascial release therapy, the therapist applies light pressure by hand to find myofascial areas that feel stiff instead of elastic and movable. These stiff areas, or trigger points, are thought to limit muscle and joint movements, which can play a part in widespread muscle pain.
  Interventions: Diagnostic Test: Myofascial Release Technique
- Ultrasound Therap (Experimental): Ultrasound physical therapy is a branch of ultrasound, alongside diagnostic ultrasound and pregnancy imaging. It's used to detect and treat various musculoskeletal issues you may have including pain, tissue injury, and muscle spasms
  Interventions: Other: Ultrasound Therapy

INTERVENTIONS:
Diagnostic Test: Myofascial Release Technique — myofascial release therapy, the therapist applies light pressure by hand to find myofascial areas that feel stiff instead of elastic and movable. These stiff areas, or trigger points, are thought to limit muscle and joint movements, which can play a part in widespread muscle pain.
  Arms: Myofascial Release Technique
Other: Ultrasound Therapy — Ultrasound physical therapy is a branch of ultrasound, alongside diagnostic ultrasound and pregnancy imaging. It's used to detect and treat various musculoskeletal issues you may have including pain, tissue injury, and muscle spasms
  Arms: Ultrasound Therap

SUMMARY:
Low back pain is common problem the purpose of this research will be to determine the comparison of ultrasound therapy and myofascial release technique for treatment of low back pain in adults.

DETAILED DESCRIPTION:
Low back pain is common problem the purpose of this research will be to determine the comparison of ultrasound therapy and myofascial release technique for treatment of low back pain in adults. To increase lumbar spine range of motion chest wall mobility and flexibility, reduction in level of lumbar disability

ELIGIBILITY:
Inclusion Criteria:

* Both male and female
* between age of 18 and 60 reported with chronic low back pain (lasting more than 3 months)

Exclusion Criteria:

* unresponsive psychologically disturbed patient
* people under 18
* Following coexisting conditions cancer, diabetes, pregnancy, cardiovascular system, gynecological disease.
* Neurological conditions, spine injury contraindicated to MFR treatment (infectious disease, viral and bacterial infections, active malignant disease, aneurysm
* Arthrodesis

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-07-10 (Actual)

PRIMARY OUTCOMES:
Modified Oswestry disability index | 6 Months
  Oswestry Disability Index [ODI] (an outcome measure that was designed to assess function in activities of daily living for those with acute or chronic back pain)

CONTACTS AND LOCATIONS:
Overall Officials: Abdul Wahab, Study Chair — Superior Uni
Locations (1):
- Azra Naheed Medical College, Superior University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No